

### East Midlands - Leicester South Research Ethics Committee

The Old Chapel Royal Standard Place Nottingham NG1 6FS

Please note: This is the favourable opinion of the REC only and does not allow you to start your study at NHS sites in England until you receive HRA Approval

02 May 2018

Dr Sancho Rodriguez-Villar Consultant in Intensive Care Medicine Kings College NHS Trust Denmark Hill Denmark Hill, Brixton, London SE5 9RS

## Dear Dr Rodriguez-Villar

| Study title: | The impact of systemic pH on cardiac function and clinical outcome in the critically ill patient |
|---|---|
| REC reference: | 18/EM/0138 |
| Protocol number: | N/A |
| IRAS project ID: | 227870 |

The Proportionate Review Sub-committee of the East Midlands - Leicester South Research Ethics Committee reviewed the above application on 02 May 2018.

We plan to publish your research summary wording for the above study on the HRA website, together with your contact details. Publication will be no earlier than three months from the date of this favourable opinion letter. The expectation is that this information will be published for all studies that receive an ethical opinion but should you wish to provide a substitute contact point, wish to make a request to defer, or require further information, please contact <a href="mailto:hra.studyregistration@nhs.net">hra.studyregistration@nhs.net</a> outlining the reasons for your request. Under very limited circumstances (e.g. for student research which has received an unfavourable opinion), it may be possible to grant an exemption to the publication of the study.



## **Ethical opinion**

On behalf of the Committee, the sub-committee gave a favourable ethical opinion of the above research on the basis described in the application form, protocol and supporting documentation, subject to the conditions specified below.

#### Conditions of the favourable opinion

The REC favourable opinion is subject to the following conditions being met prior to the start of the study.

Management permission must be obtained from each host organisation prior to the start of the study at the site concerned.

Management permission should be sought from all NHS organisations involved in the study in accordance with NHS research governance arrangements. Each NHS organisation must confirm through the signing of agreements and/or other documents that it has given permission for the research to proceed (except where explicitly specified otherwise).

Guidance on applying for HRA and HCRW Approval (England and Wales)/ NHS permission for research is available in the Integrated Research Application System, <a href="http://www.rdforum.nhs.uk">www.hra.nhs.uk</a> or at <a href="http://www.rdforum.nhs.uk">http://www.rdforum.nhs.uk</a>.

Where a NHS organisation's role in the study is limited to identifying and referring potential participants to research sites ("participant identification centre"), guidance should be sought from the R&D office on the information it requires to give permission for this activity.

For non-NHS sites, site management permission should be obtained in accordance with the procedures of the relevant host organisation.

Sponsors are not required to notify the Committee of management permissions from host organisations.

#### Registration of Clinical Trials

All clinical trials (defined as the first four categories on the IRAS filter page) must be registered on a publically accessible database. This should be before the first participant is recruited but no later than 6 weeks after recruitment of the first participant.

There is no requirement to separately notify the REC but you should do so at the earliest opportunity e.g. when submitting an amendment. We will audit the registration details as part of the annual progress reporting process.

To ensure transparency in research, we strongly recommend that all research is registered but for non-clinical trials this is not currently mandatory.



If a sponsor wishes to request a deferral for study registration within the required timeframe, they should contact <a href="https://doi.org/10.21/10.1016/j.net">https://doi.org/10.21/10.1016/j.net</a>. The expectation is that all clinical trials will be registered, however, in exceptional circumstances non registration may be permissible with prior agreement from the HRA. Guidance on where to register is provided on the HRA website.

It is the responsibility of the sponsor to ensure that all the conditions are complied with before the start of the study or its initiation at a particular site (as applicable).

#### Ethical review of research sites

The favourable opinion applies to all NHS sites taking part in the study, subject to management permission being obtained from the NHS/HSC R&D office prior to the start of the study (see "Conditions of the favourable opinion").

#### Summary of discussion at the meeting

### Social or scientific value; scientific design and conduct of the study

The Sub-Committee noted section 2a of the IRAS application indicates the study will use identifiable data, whereas the section 4b states the research is limited to use of previously collected, non-identifiable information. The Sub-Committee noted all data will be collected by the direct care team and anonymised before sending for statistical analysis, and agreed the study meets the 'no material ethical issues' criteria.

#### **Approved documents**

The documents reviewed and approved were:

| Document | Version | Date |
|---|---|---|
| IRAS Application Form [IRAS_Form_18042018] | | 18 April 2018 |
| IRAS Checklist XML [Checklist_18042018] | | 18 April 2018 |
| Research protocol or project proposal [227870 pH in critically ill patients- Protocol- 25.01.2018] | 1.0 | 25 January 2018 |
| Summary CV for Chief Investigator (CI) [Sancho Rodriguez-Villar CV] | | 22 July 2017 |

#### **Membership of the Proportionate Review Sub-Committee**

The members of the Sub-Committee who took part in the review are listed on the attached sheet.

## Statement of compliance

The Committee is constituted in accordance with the Governance Arrangements for Research Ethics Committees and complies fully with the Standard Operating Procedures for Research Ethics Committees in the UK.



#### After ethical review

## Reporting requirements

The attached document "After ethical review – guidance for researchers" gives detailed guidance on reporting requirements for studies with a favourable opinion, including:

- Notifying substantial amendments
- · Adding new sites and investigators
- Notification of serious breaches of the protocol
- Progress and safety reports
- Notifying the end of the study

The HRA website also provides guidance on these topics, which is updated in the light of changes in reporting requirements or procedures.

#### User Feedback

The Health Research Authority is continually striving to provide a high quality service to all applicants and sponsors. You are invited to give your view of the service you have received and the application procedure. If you wish to make your views known please use the feedback form available on the HRA website:

http://www.hra.nhs.uk/about-the-hra/governance/guality-assurance/

#### **HRA Training**

We are pleased to welcome researchers and R&D staff at our training days – see details at <a href="http://www.hra.nhs.uk/hra-training/">http://www.hra.nhs.uk/hra-training/</a>

With the Committee's best wishes for the success of this project.



## 18/EM/0138

Please quote this number on all correspondence

Yours sincerely

huallace

pp

Mr John Aldridge

Chair

Email: NRESCommittee.EastMidlands-LeicesterSouth@nhs.net

Enclosures: List of names and professions of members who took part in the review

"After ethical review – guidance for researchers"

Copy to: Miss Liba Stones, The R&I Office, King's College Hospital NHS

Foundation Trust



## **East Midlands - Leicester South Research Ethics Committee**

# Attendance at PRS Sub-Committee of the REC meeting on 02 May 2018

## **Committee Members:**

| Name | Profession | Present | Notes |
|---|---|---|---|
| Mr John Aldridge (Chair) | Retired Senior Lecturer in Nursing | Yes | |
| Ms Elizabeth Gibbons | Senior Research<br>Scientist | Yes | |
| Mrs Jill Marshall | Retired Training and Development Manager | Yes | |

## Also in attendance:

| Name | Position (or reason for attending) |
|----------------------|------------------------------------|
| Miss Lindsey Wallace | REC Manager |